CLINICAL TRIAL: NCT05901467
Title: Recall by Genotype: Neuropeptide Stimulation
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study team no longer has access to GnRH. The study has been altered to account for this change and is no longer a clinical trial.
Sponsor: Stephanie B. Seminara, MD (Other)
Responsible Party: Sponsor-Investigator, Stephanie B. Seminara, MD, Chief, Reproductive Endocrine Unit; Professor of Medicine, Harvard Medical School; Director, MGH Harvard Center for Reproductive Medicine, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 326733; P50HD104224 (NIH)
Record Dates: First submitted 2023-05-31; First posted 2023-06-13 (Actual); Results first posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Reproductive Disorder
Keywords: reproductive disorders; kisspeptin; infertility; GnRH
MeSH Terms: conditions — Infertility | interventions — Gonadotropin-Releasing Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- kisspeptin, GnRH (Experimental): IV administration of kisspeptin 112-121; one bolus. IV administration of GnRH; one bolus.
  Interventions: Drug: kisspeptin 112-121; Drug: GnRH

INTERVENTIONS:
Drug: kisspeptin 112-121 — One IV bolus of kisspeptin 112-121
  Other Names: metastin 45-54
Drug: GnRH — One IV bolus of gonadotropin-releasing hormone
  Other Names: gonadotropin-releasing hormone

SUMMARY:
The objective of this protocol is to assess response to kisspeptin and gonadotropin-releasing hormone (GnRH) stimulation testing as well as the baseline patterns of luteinizing hormone (LH) secretion in individuals who carry variants in genes related to infertility.

DETAILED DESCRIPTION:
Assignment: All study subjects will undergo the same interventions. Individuals at high risk for infertility (i.e., carry variants in genes related to infertility) will be compared to controls (i.e., those who do not carry variants in genes related to infertility).

Delivery of Interventions:

* Prior to the inpatient study visit, the subjects will undergo a review of their medical history, physical exam, and screening laboratories.
* On the day of the study, the subjects will have an intravenous (IV) line placed and

  * Undergo up to q10 min blood sampling x 12 hours
  * Receive a single kisspeptin IV bolus at hour 8
  * Receive a single GnRH IV bolus at hour 11

ELIGIBILITY:
Inclusion Criteria:

* No prescription medications that could interfere with hypothalamic reproductive function
* No illicit drug use
* No excessive alcohol consumption (more than 10 drinks/week)
* No history of an allergic medication reaction requiring emergency medical care
* Normal blood pressure reading (systolic blood pressure < 140 mm Hg, diastolic < 90 mm Hg)
* White blood cell, platelet counts, prolactin, and thyroid-stimulating hormone (TSH) between 90% of the lower limit and 110% of the upper limit of the reference range
* Normal hemoglobin
* Blood urea nitrogen (BUN), creatinine not elevated
* Aspartate aminotransferase (AST), alanine aminotransferase (ALT) within 3 times upper limit of normal
* Enrolled in the Partners HealthCare Biobank and genotypically characterized
* For women

  * No oral contraceptives for at least 1 month
  * No contraceptive implants for at least 3 months
  * Not breastfeeding and not pregnant
  * Negative serum human chorionic gonadotropin (hCG) pregnancy test at the time of screening (additional urine pregnancy test will be conducted prior to drug administration)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2023-10-20 (Actual); Primary Completion 2024-05-29 (Actual); Study Completion 2024-05-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie B Seminara, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Boston area. 16 participants were consented and screened for eligibility between 10/2023 and 4/2024.
Pre-assignment Details: There was no washout or run-in period. 4 individuals were found to be ineligible by criteria.
Period: Overall Study
Arm/Group | kisspeptin, GnRH
Started | 16
Completed | 0
Not Completed | 16

BASELINE CHARACTERISTICS:
Arm/Group | Kisspeptin, GnRH
Number analyzed (Participants) | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 12
  More than one race | 0
  Unknown or Not Reported | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 0

OUTCOME MEASURES:

1. Primary Outcome: Endogenous LH Pulse Amplitude
Description: Average amplitude of LH pulses at baseline
Time Frame: Hours 0-8
Population: No participants underwent the intervention. This trial was terminated because the study team no longer had access to the study drugs.
Measure: Mean (Standard Deviation); unit: mIU/mL
Arm/Group | kisspeptin, GnRH
Number analyzed (Participants) | 0

2. Primary Outcome: Kisspeptin-induced LH Pulse Amplitude
Description: Amplitude of LH pulse in response to kisspeptin
Time Frame: Hours 8-11
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mIU/mL
Arm/Group | kisspeptin, GnRH
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From time of study consent until removal from study participation (approximately 2 months).
Description: All participants were asked about new health symptoms at each visit.
Arm/Group | kisspeptin, GnRH
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 1/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | kisspeptin, GnRH (N=16)
Upper respiratory infection (Infections and infestations) | 1 — The primary healthcare team of the participant informed the study team of this adverse event. The event was determined to be grade 1 and unrelated to study interventions.

LIMITATIONS AND CAVEATS:
No participants underwent the intervention. This trial was terminated because the study team no longer had access to the study drugs.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-10-31): https://cdn.clinicaltrials.gov/large-docs/67/NCT05901467/Prot_SAP_000.pdf